CLINICAL TRIAL: NCT03720405
Title: Measurement of the Distance Between the Corresponding Anatomical Landmarks in the Thoracic Cavity and the Incisors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2018-85
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Pulmonary Resection
Keywords: pulmonary resection; Esophageal segmentation; Regression equation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients who agree to receive pneumonectomy will be arranged to measure the distance from the incisors to the corresponding anatomical landmarks, including the cardia, the inferior pulmonary vein, the carina, the azygos vein, the lower edge of the aortic arch, the upper edge of the aortic arch, and the cupula of pleura through " fiber measurement method within nasogastric tube " . After building regression equations with the above data, the distance from the incisors to these corresponding anatomical landmarks could be inferred by means of indexes including height and so on.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing thoracic operation(such as radical lung cancer resection, pulmonary lobectomy, pulmonary segmentectomy, etc.) under endotracheal anesthesia ,which can expose the corresponding anatomical landmarks;
* Patients undergoing nasogastric intubation due to their condition.

Exclusion Criteria:

* Patients with diseased or deformed esophagus;
* Patients with obvious thoracic deformity, spinal deformity or dysplasia;
* Patients whose thoracic anatomical landmarks can not be exposed or exposed clearly during operation;
* Patients who do not agree to be measured.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient from Department of Thoracic Surgery, Southern Hospital of Southern Medical University.
Sampling Method: Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
the distance from the incisors to the corresponding anatomical landmarks | 1 hour
  The distance from the thoracic anatomical landmarks (the lower edge of the cardia, the inferior pulmonary vein, the condyle, the lower edge of the azygous vein, the lower edge of the aortic arch, the upper edge of the aortic arch, and the pleural apex) to the incisors.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guandong, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
The results of distance measurement of each individual participant.

REFERENCES:
- [Background] Japan Esophageal Society. Japanese Classification of Esophageal Cancer, 11th Edition: part I. Esophagus. 2017;14(1):1-36. doi: 10.1007/s10388-016-0551-7. Epub 2016 Nov 10. No abstract available. PMID 28111535
- [Background] Rice TW, Ishwaran H, Ferguson MK, Blackstone EH, Goldstraw P. Cancer of the Esophagus and Esophagogastric Junction: An Eighth Edition Staging Primer. J Thorac Oncol. 2017 Jan;12(1):36-42. doi: 10.1016/j.jtho.2016.10.016. Epub 2016 Oct 31. PMID 27810391
- [Background] Biere SS, van Berge Henegouwen MI, Maas KW, Bonavina L, Rosman C, Garcia JR, Gisbertz SS, Klinkenbijl JH, Hollmann MW, de Lange ES, Bonjer HJ, van der Peet DL, Cuesta MA. Minimally invasive versus open oesophagectomy for patients with oesophageal cancer: a multicentre, open-label, randomised controlled trial. Lancet. 2012 May 19;379(9829):1887-92. doi: 10.1016/S0140-6736(12)60516-9. Epub 2012 May 1. PMID 22552194
- [Background] Lagergren J, Smyth E, Cunningham D, Lagergren P. Oesophageal cancer. Lancet. 2017 Nov 25;390(10110):2383-2396. doi: 10.1016/S0140-6736(17)31462-9. Epub 2017 Jun 22. PMID 28648400
- [Background] Javidfar J, Speicher PJ, Hartwig MG, D'Amico TA, Berry MF. Impact of Positive Margins on Survival in Patients Undergoing Esophagogastrectomy for Esophageal Cancer. Ann Thorac Surg. 2016 Mar;101(3):1060-7. doi: 10.1016/j.athoracsur.2015.09.005. Epub 2015 Nov 11. PMID 26576752
- [Background] Markar SR, Gronnier C, Duhamel A, Pasquer A, Thereaux J, Chalret du Rieu M, Lefevre JH, Turner K, Luc G, Mariette C; FREGAT Working Group-FRENCH-AFC. Significance of Microscopically Incomplete Resection Margin After Esophagectomy for Esophageal Cancer. Ann Surg. 2016 Apr;263(4):712-8. doi: 10.1097/SLA.0000000000001325. PMID 26135681
- [Background] Gilbert S, Martel AB, Seely AJ, Maziak DE, Shamji FM, Sundaresan SR, Villeneuve PJ. Prognostic significance of a positive radial margin after esophageal cancer resection. J Thorac Cardiovasc Surg. 2015 Feb;149(2):548-55; discussion 555. doi: 10.1016/j.jtcvs.2014.10.040. Epub 2014 Oct 14. PMID 25454924
- [Background] Chan DS, Reid TD, Howell I, Lewis WG. Systematic review and meta-analysis of the influence of circumferential resection margin involvement on survival in patients with operable oesophageal cancer. Br J Surg. 2013 Mar;100(4):456-64. doi: 10.1002/bjs.9015. Epub 2013 Jan 14. PMID 23319427
- [Background] Okada N, Fujii S, Fujita T, Kanamori J, Kojima T, Hayashi R, Daiko H. The prognostic significance of the positive circumferential resection margin in pathologic T3 squamous cell carcinoma of the esophagus with or without neoadjuvant chemotherapy. Surgery. 2016 Feb;159(2):441-50. doi: 10.1016/j.surg.2015.06.044. Epub 2015 Sep 19. PMID 26391150
- [Background] Wu J, Chen QX, Teng LS, Krasna MJ. Prognostic significance of positive circumferential resection margin in esophageal cancer: a systematic review and meta-analysis. Ann Thorac Surg. 2014 Feb;97(2):446-53. doi: 10.1016/j.athoracsur.2013.10.043. Epub 2013 Dec 21. PMID 24365211
- [Background] Korn O, Csendes A, Burdiles P, Braghetto I, Sagastume H, Biagini L. Length of the esophagus in patients with gastroesophageal reflux disease and Barrett's esophagus compared to controls. Surgery. 2003 Apr;133(4):358-63. doi: 10.1067/msy.2003.117. PMID 12717351